CLINICAL TRIAL: NCT03853135
Title: Assessment of Endocan Serum Levels in Patients With Behcet Disease: Relation to Clinical Parameters and Disease Status
Brief Title: Assessment of Endocan Serum Levels in Patients With Behcet Disease
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Waleed Ahmed Salaheldeen Hassan, Assistant professor, Benha University
Other Study IDs: BenhaU22019
Record Dates: First submitted 2019-02-22; First posted 2019-02-25 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Behçet
Keywords: Behçet disease; endocan
MeSH Terms: conditions — Behcet Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Behçet group: Forty two patients diagnosed to have Behçet disease fulfilling the International Study Group Criteria for Behçet disease in whom measurement of serum endocan levels will be performed.
  Interventions: Diagnostic Test: measurement of serum endocan
- control group: including 42 age and sex matching healthy volunteers as control group in whom measurement of serum endocan levels will be performed.
  Interventions: Diagnostic Test: measurement of serum endocan

INTERVENTIONS:
Diagnostic Test: measurement of serum endocan — measurement of serum levels of endocan
  Other Names: endothelial cell-specific molecule 1

SUMMARY:
The aim of our study was to assess serum endocan levels in patients with Behcet disease and to correlate it with various disease clinical and laboratory parameters of disease activity as well as carotid intima media thickness.

DETAILED DESCRIPTION:
This study will be carried out on two groups:

• Group (I): Forty two patients diagnosed to have Behcets disease fulfilling the International Criteria for BD .

Group (II): including 42 age and sex matching healthy volunteers as control group.

(A) Clinical evaluation

1. Complete history taking.
2. Thorough clinical examination including opthalmologic evaluation .
3. Disease activity using The Behcet's disease current activity form (BD-DAF) . (B) Laboratory assessment:

All patients will be subjected to the following measurements:

1. ESR
2. CRP
3. CBC
4. liver and kidney function tests

d) Serum Endocan level e)triglycrides f) cholestrol C) carotid intima media thickness

ELIGIBILITY:
Inclusion Criteria:

* patients with Behcets disease fulfilling the International Criteria for BD .

Exclusion Criteria:

* infection
* malignancy
* other connective tissue disease
* chronic liver disease
* chronic kidney disease
* Diabetes mellitus
* hypertension
* hyperlipidemia

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will be carried out on two groups:
  • Group (I): Forty two patients diagnosed to have Behcets disease fulfilling the International Criteria for BD .
  Group (II): including 42 age and sex matching healthy volunteers as control group.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
the Behcet's disease current activity form (BDCAF) | : through study completion, an average of 6 months
  One point is given to the presence of different organ involvement over the 4 weeks prior to assessment as follows: headache, mouth ulcers, genital ulcers, skin lesions , joint involvement , gastrointestinal symptoms , eye involvement , nervous system involvement , and major vessel involvement.The total score will be out of 12 and higher score indicates worse outcome. we will assess the relation between serum endocan level and BDCAF
Erythrocyte sedimentation rate (ESR) | : through study completion, an average of 6 months
  ESR measured in mm/1st hour by westergren method. we will assess the relation between serum endocan level and ESR
C reactive protein (CRP) | : through study completion, an average of 6 months
  CRP measured in mg/L using nephlometry. we will assess the relation between serum endocan level and CRP
carotid intima media thickness | : through study completion, an average of 6 months
  Color Doppler ultrasonography was performed for both common carotid arteries in a longitudinal orientation and measured with millimeter

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Hassan, MD, Principal Investigator — Benha university- Qaluibya- Egypt
Locations (1):
- Benha University Hospital, Banhā, Qalyubia Governorate, Egypt